CLINICAL TRIAL: NCT02285127
Title: Short Versus Long Cephalomedullary Nailing of Pertrochanteric Hip Fractures: A Randomized Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen A. Sems, Assistant Professor of Orthopedics, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-002490
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Pertrochanteric Hip Fracture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short nail implant (Active Comparator): used to treat pertrochanteric fractures
  Interventions: Procedure: Short versus long cephalomedullary Intramedullary nail
- Long nail implant (Active Comparator): used to treat pertrochanteric fractures
  Interventions: Procedure: Short versus long cephalomedullary Intramedullary nail

INTERVENTIONS:
Procedure: Short versus long cephalomedullary Intramedullary nail — Biomet Affixus Short and Long hip fracture nail. Stryker Gamma Short and Long hip fracture nail.

SUMMARY:
Is there a functional outcome difference when treating pertrochanteric fractures with a short or long cephalomedullary nail?

ELIGIBILITY:
Inclusion criteria

* AO/OTA fracture classification 31(A-B) (1-3).
* Age greater than 18 years old.

Exclusion Criteria

-Less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-11; Primary Completion 2018-05-01 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
SF (short form)-36 | 3 months

SECONDARY OUTCOMES:
Harris Hip Score | 3 months

OTHER OUTCOMES:
Reoperation | within 1 year
Mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Sems, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials